CLINICAL TRIAL: NCT00718159
Title: Phase 1 Study of LY573636-sodium in Patients With Essential Thrombocythemia and Acute Myeloid Leukemia
Brief Title: Study of LY573636-sodium in Essential Thrombocythemia and Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12266; H8K-MC-JZAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Acute Myeloid Leukemia; Essential Thrombocythemia
Keywords: Acute Myeloid Leukemia; Myeloid Leukemia; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Thrombocythemia, Essential; Leukemia, Myeloid; Recurrence | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY573636 (Experimental)
  Interventions: Drug: LY573636-sodium

INTERVENTIONS:
Drug: LY573636-sodium — Individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Dosing will be done on Day 1 of a 35-day cycle for acute myeloid leukemia (AML) and Day 1 of a 28-day cycle for essential thrombocythemia (ET) for at least one cycle. A participant may have additional cycles of LY573636 if he or she is receiving benefit from the study drug and does not fulfill any of the criteria for study discontinuation.
  Other Names: LY573636

SUMMARY:
The purpose of this study is to determine a safe dose of LY573636-sodium to be given to patients with acute myeloid leukemia and to determine any side effects that may be associated with LY573636-sodium in this patient population. Efficacy measures will also be used to assess the activity of LY573636-sodium in acute myeloid leukemia and essential thrombocythemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a diagnosis of either essential thrombocythemia or acute myeloid leukemia that is relapsed or refractory to at least one prior standard treatment. If participants have acute promyelocytic leukemia, they must be resistant and/or intolerant of both all trans retinoic acid (ATRA) and arsenic trioxide.
* Are at least 18 years of age.
* Have given written informed consent approved by Lilly and the ethical review board (ERB)/institutional review board (IRB) governing the site.
* Must have adequate hepatic and renal function.
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, immunotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 21 days for myelosuppressive agents (such as cytarabine, daunorubicin, and gemtuzumab ozogamicin) or 14 days for non-myelosuppressive agents prior to receiving study drug and recovered from the acute effects of therapy. Hydroxyurea used to control peripheral blood blast count is permitted within these respective periods, but it must be stopped at least 24 hours before study drug administration.
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drug.
* Females of child bearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug.
* Have a serum albumin level greater than equal to 3.0 grams/deciliter (g/L), less than or equal to 72 hour prior to dosing with LY573636-sodium.

Exclusion Criteria:

* Have received treatment with a drug that has not received regulatory approval for any indication within 14 or 21 days of the initial dose of study drug for a non-myelosuppressive or myelosuppressive agent, respectively.
* Participants with myeloproliferative disorders (for example, chronic myeloid leukemia (CML), polycythemia vera and primary myelofibrosis) other than essential thrombocythemia.
* Have received an autologous or allogenic stem cell transplant within 75 days of the initial dose of study drug for the dose escalation phase or within 60 days of the initial dose of study drug for the dose confirmation phase. Recipients of an allogeneic stem cell transplant must have discontinued immunosuppressive therapy at least 24 hours before study drug administration with no more than Grade 1 acute graft-versus-host disease.
* Have previously completed or withdrawn from this study or any other study investigating LY573636 sodium.
* Have serious preexisting medical conditions that in the opinion of the investigator would preclude participation in this study.
* Have serious concomitant disorders, including active bacterial, fungal, or viral infection, incompatible with the study.
* Have a second primary malignancy that could affect interpretation of results.
* Have a known coagulopathy or bleeding disorder, other than leukemic related thrombocytopenia. Participants with severe or life-threatening bleeding refractory to platelet transfusions are also excluded from this study.
* Major surgery within 4 weeks of study enrollment.
* Are receiving warfarin (Coumadin).
* Females who are pregnant or breast feeding.
* Have known positive results of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBSAg) or hepatitis C antibodies (HCAb).
* Have received treatment within 28 days of the initial dose of study drug with an experimental agent for noncancerous indications that has not received regulatory approval for any indication.
* Participants receiving amiodarone, quinidine, propofol, or clozapine.
* Participants receiving treatment with strong or moderate inhibitors of cytochrome P450 (CYP)2C19, including proton-pump inhibitors (PPIs). Esomeprazole or pantoprazole are allowed if not administered within 72 hours before or after LY573636 administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon -Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment. All participants who received at least 1 dose of study drug were considered to have completed the study.
Groups:
- Cmax 250 μg/mL (AML): Participants diagnosed with acute myeloid leukemia (AML) dosed: LY573636 targeting a maximum concentration (Cmax) of 250 micrograms per milliliter (μg/mL) as a 24-hour infusion on Day 1 of a 35-day cycle.
- Cmax 300 μg/mL (AML): Participants diagnosed with AML dosed: LY573636 targeting a Cmax of 300 μg/mL as a 24-hour infusion on Day 1 of a 35-day cycle.
- Cmax 350 μg/mL (AML): Participants diagnosed with AML dosed: LY573636 targeting a Cmax of 350 μg/mL as a 24-hour infusion on Day 1 of a 35-day cycle.
- Cmax 400 μg/mL (AML): Participants diagnosed with AML dosed: LY573636 targeting a Cmax of 400 μg/mL as a 24-hour infusion on Day 1 of a 35-day cycle.
- AUCalb 5500 µg*hr/mL (AML): Participants diagnosed with AML dosed: LY573636 targeting an albumin-corrected exposure (AUCalb) 5500 micrograms*hour per milliliter (µg*hr/mL) as a 2-hour infusion on Day 1 of a 35-day cycle.
- AUCalb 7000 µg*hr/mL (AML): Participants diagnosed with AML dosed: LY573636 targeting an AUCalb 7000 µg*hr/mL as a 2-hour infusion on Day 1 of a 35-day cycle.
- AUCalb 5500 µg*hr/mL (ET): Participants diagnosed with essential thrombocythemia (ET) dosed: LY573636 targeting an AUCalb 5500 µg*hr/mL as a 2-hour infusion on Day 1 of a 28-day cycle.
Period: Overall Study
Arm/Group | Cmax 250 μg/mL (AML) | Cmax 300 μg/mL (AML) | Cmax 350 μg/mL (AML) | Cmax 400 μg/mL (AML) | AUCalb 5500 µg*hr/mL (AML) | AUCalb 7000 µg*hr/mL (AML) | AUCalb 5500 µg*hr/mL (ET)
Started | 3 | 3 | 3 | 4 | 8 | 1 | 1
Received at Least 1 Dose of Study Drug | 3 | 3 | 3 | 4 | 8 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 4 | 8 | 1 | 1
Not completed — Progressive Disease | 3 | 3 | 2 | 0 | 6 | 0 | 0
Not completed — Death due to Adverse Event | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Death due to Study Drug Toxicity | 0 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Investigator Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cmax 250 μg/mL (AML) | Cmax 300 μg/mL (AML) | Cmax 350 μg/mL (AML) | Cmax 400 μg/mL (AML) | AUCalb 5500 µg*hr/mL (AML) | AUCalb 7000 µg*hr/mL (AML) | AUCalb 5500 µg*hr/mL (ET) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 8 | 1 | 1 | 23
Age, Continuous [Median (Full Range); unit: years] | 55.22 [55.16 to 76.21] | 52.48 [49.40 to 58.36] | 66.62 [54.69 to 75.70] | 55.46 [50.14 to 64.83] | 58.57 [24.16 to 82.19] | 81.19 [NA to NA] — Only one participant, therefore range is not calculable. | 65.09 [NA to NA] — Only one participant, therefore range is not calculable. | 56.86 [24.16 to 82.19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 4 | 0 | 1 | 14
  Male | 1 | 1 | 1 | 1 | 4 | 1 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Caucasian | 3 | 3 | 3 | 2 | 6 | 1 | 1 | 19
  Race: East Asian | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Race: Missing | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 4 | 8 | 1 | 1 | 23

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose of LY573636-Sodium in Participants With Relapsed or Refractory Acute Myeloid Leukemia (AML) and Essential Thrombocythemia (ET)
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD). MTD is the highest dose at which no more than 1 of 6 participants experienced a dose-limiting toxicity (DLT) and level immediately below that which had ≥2 instances of DLT. A DLT is an adverse event (AE) observed during the first cycle of treatment that is believed to be related to LY573636 and fulfills any of the following: ET only , Common Terminology Criteria for AE (CTCAE, Version 3.0) Grade (Gr) 4 hematologic toxicity for ≥3 days; For all, ≥Gr 3 nonhematological toxicity except for nausea/vomiting or diarrhea unless it fits the next criteria; ≥Gr 3 nausea, vomiting, or diarrhea that persists >7 days despite maximal treatment; Gr 3 electrolyte disturbances that persist despite maximal measures; DLT can be declared if a participant experienced increasing toxicity during treatment. The primary outcome measure was not analyzed because the enrollment was stopped early before MTD was reached.
Time Frame: Predose up to 35 days postdose in Cycle 1
Population: No participants were analyzed since the MTD was not reached.
Arm/Group | Cmax 250 μg/mL (AML) | Cmax 300 μg/mL (AML) | Cmax 350 μg/mL (AML) | Cmax 400 μg/mL (AML) | AUCalb 5500 µg*hr/mL (AML) | AUCalb 7000 µg*hr/mL (AML) | AUCalb 5500 µg*hr/mL (ET)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics Area Under the Curve(AUC) of LY573636 Above the Albumin-Corrected Threshold (AUCalb)
Description: LY573636 has been found to be highly bound to albumin. AUCalb is a surrogate measure of exposure to unbound (free) LY573636.
  PK sample is withdrawn at any time on days 8,14,15,21,28.
Time Frame: Predose,1h,2h,4h, 8d,14d,15d,21d,28d post dose
Population: Participants who received the study drug and had pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*hr/mL)
Groups:
- LY573636: LY573636 dose was based on an albumin-corrected exposure (AUCalb) to target a specific exposure range. Intravenous dosing is done on Day 1 of Cycle 1. Data are pooled together from all treatment groups.
Arm/Group | LY573636
Number analyzed (Participants) | 23
micrograms*hour/milliliter (µg*hr/mL) | 6911 (86.8)

3. Secondary Outcome: Number of Participants With Bone Marrow (BM) Response
Description: The International Working Group's revised recommendations were used to assess response in acute myeloid leukemia (AML): complete response (CR) is <5% blasts in BM and with a cell count ≥200 cells in BM, and with peripheral blood platelets ≥100x10⁹/liter (L) and absolute neutrophils ≥1x10⁹/L; CR with incomplete blood count recovery is defined as CRi; partial response (PR) is ≥5% blasts in BM but with ≥50% reduction in blast count. Number of responders for AML = CR+PR+ CRi. Result of a European Leukemia Net consensus conference was used to assess response in essential thrombocythemia (ET). CR is platelets ≤400x10⁹/L in peripheral blood, no disease-related symptoms, normal spleen size and white blood cells ≤10x10⁹/L in peripheral blood; PR has platelets ≤600x10⁹/L in peripheral blood or decrease > 50% from baseline but does not meet CR criteria. Number of responders for ET = CR+PR.
Time Frame: Baseline to measured progressive disease up to 70 days
Population: All participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cmax 250 μg/mL (AML) | Cmax 300 μg/mL (AML) | Cmax 350 μg/mL (AML) | Cmax 400 μg/mL (AML) | AUCalb 5500 µg*hr/mL (AML) | AUCalb 7000 µg*hr/mL (AML) | AUCalb 5500 µg*hr/mL (ET)
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 8 | 1 | 1
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetics: Concentration Maximum (Cmax) of LY573636
Description: PK sample is withdrawn at any time on days 8,14,15,21,28.
Time Frame: Predose,1h,2h,4h, 8d,14d,15d,21d,28d post dose
Population: Participants who received the study drug and had pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | LY573636
Number analyzed (Participants) | 23
micrograms per milliliter (µg/mL) | 317 (21.0)

ADVERSE EVENTS:
Groups:
- AUCalb 5500 µg*hr/mL (AML and ET): Participants diagnosed with AML dosed: LY573636 targeting an albumin-corrected exposure (AUCalb) 5500 micrograms*hour per milliliter (µg*hr/mL) as a 2-hour infusion on Day 1 of a 35-day cycle.
  Participants diagnosed with essential thrombocythemia (ET) dosed: LY573636 targeting an AUCalb 5500 µg*hr/mL as a 2-hour infusion on Day 1 of a 28-day cycle.
Arm/Group | Cmax 250 μg/mL (AML) | Cmax 300 μg/mL (AML) | Cmax 350 μg/mL (AML) | Cmax 400 μg/mL (AML) | AUCalb 5500 µg*hr/mL (AML and ET) | AUCalb 7000 µg*hr/mL (AML)
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 1/3 | 4/4 | 6/9 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 9/9 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cmax 250 μg/mL (AML) (N=3) | Cmax 300 μg/mL (AML) (N=3) | Cmax 350 μg/mL (AML) (N=3) | Cmax 400 μg/mL (AML) (N=4) | AUCalb 5500 µg*hr/mL (AML and ET) (N=9) | AUCalb 7000 µg*hr/mL (AML) (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Resulted in a death in the Cmax 400 μg/mL (AML) arm
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Resulted in 2 deaths in the Cmax 400 μg/mL (AML) arm
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Resulted in a death in the Cmax 350 μg/mL (AML) arm and in the Cmax 400 μg/mL
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Resulted in a death in the AUCalb 5500 µg*hr/mL (AML) arm
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Resulted in a death in the AUCalb 5500 µg*hr/mL (AML) arm
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cmax 250 μg/mL (AML) (N=3) | Cmax 300 μg/mL (AML) (N=3) | Cmax 350 μg/mL (AML) (N=3) | Cmax 400 μg/mL (AML) (N=4) | AUCalb 5500 µg*hr/mL (AML and ET) (N=9) | AUCalb 7000 µg*hr/mL (AML) (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 2 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Inflammatory pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Therapeutic response unexpected (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 4 (5) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0/2 (0) | 0/2 (0) | 0/2 (0) | 1/3 (1) | 0/5 (0) | 0/0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary outcome measure in this trial was not reached because the enrollment was stopped early before the maximum tolerated dose was reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days